CLINICAL TRIAL: NCT00701285
Title: A Prospective, Randomized, Two Group Comparison Study to Evaluate the Effect of Statin on Heart Function in Patients With Chronic Ischemic Heart Failure.
Brief Title: South Korean Pitavastatin Heart Failure Study
Acronym: SAPHIRE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: JW Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CWP-PTV-703
Record Dates: First submitted 2008-06-17; First posted 2008-06-19 (Estimated); Last update posted 2014-05-14 (Estimated); Status verified 2014-05

CONDITIONS: Chronic Heart Failure
Keywords: heart failure; pitavastatin; pravastatin; statin
MeSH Terms: conditions — Heart Failure | interventions — pitavastatin; Pravastatin

ARMS (2):
- 1 (Active Comparator): strong statin
  Interventions: Drug: pitavastatin
- 2 (Active Comparator): mild statin
  Interventions: Drug: pravastatin

INTERVENTIONS:
Drug: pitavastatin — pitavastatin 4mg once daily
  Arms: 1
Drug: pravastatin — pravastatin 10mg once daily
  Arms: 2

SUMMARY:
We want to evaluate the utility of statins on heart function according to potency. Patients with chronic ischemic heart failure are administered pitavastatin 4mg or pravastatin 10mg for 52 weeks. Then we evaluate the effect of pitavastatin and pravastatin primarily on rate of hospitalization for cardiovascular cause and lipid profile secondarily biomarker, echocardiography parameter, 6-minute walk, change of NYHA class distribution, cardiovascular mortality.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who accepted to enter the study by written informed consent
2. Age ≥ 30 years
3. LDL-cholesterol ≥ 70mg/dl
4. Chronic heart failure of :

   * NYHA class II ~ III
   * Ischemic etiology
   * Left ventricular ejection fraction < 45%
   * Optimal therapy for chronic heart failure and stable clinical condition over the two weeks.

Exclusion Criteria:

1. Patients who participated in other studies 3 months before enrollment
2. Statin treatment within 2 months before enrollment
3. Unstable decompensated heart failure at enrollment
4. Acute coronary syndrome or cerebral vascular disease within 3 months before enrollment
5. Coronary revascularization within 3 months before enrollment or planned at enrollment
6. Any other serious disease or condition which might effect life expectancy such as malignancy, life-threatening infectious disease.
7. Serum creatinine levels >= 3.0 mg/dl
8. AST or AST levels >=2.5 times of ULN
9. CK levels >=2 times of ULN
10. Uncontrolled hypothyroidism : TSH level >= 2 times of ULN
11. Pregnant or breastfeeding women, women who want to bearing
12. Patients who might to be unsuitable by the decision of investigators

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2008-07; Primary Completion 2013-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Rate and number of hospitalization for cardiovascular cause; Lipid profile | 52week

SECONDARY OUTCOMES:
Biomarker : BNP, hsCRP, IL-6. TNF-α | 52 week
Echocardiography : LVEF, E/A ratio, LVEDD, LVESD | 52 week
Cardiac function evaluation (NYHA class distribution, 6-minute walk test) | 52 week
Cardiovascular mortality | 52 week

CONTACTS AND LOCATIONS:
Overall Officials: Sang Hong Baek, MD, PhD, Study Chair — KangNam St. Mary's Hospital
Locations (1):
- SEOUL St. Mary's Hospital, Seoul, Seocho-Ku, South Korea

REFERENCES:
- [Derived] Lee HY, Cho HJ, Kim HY, Jeon HK, Shin JH, Kang SM, Baek SH. Effects of intensive versus mild lipid lowering by statins in patients with ischemic congestive heart failure: Korean Pitavastatin Heart Failure (SAPHIRE) study. Korean J Intern Med. 2014 Nov;29(6):754-63. doi: 10.3904/kjim.2014.29.6.754. Epub 2014 Oct 31. PMID 25378974